CLINICAL TRIAL: NCT05562154
Title: Lateral Approach Versus Anterior Approach in Total Ankle Replacement: A Randomized Clinical Trial
Brief Title: Lateral Approach Versus Anterior Approach in Total Ankle Replacement
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution and successor no longer interested in topic.
Sponsor: John Femino (Other)
Responsible Party: Sponsor-Investigator, John Femino, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202010410
Record Dates: First submitted 2022-08-25; First posted 2022-09-30 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Ankle Osteoarthritis
MeSH Terms: interventions — Arthroplasty, Replacement, Ankle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lateral Approach (Active Comparator)
  Interventions: Procedure: Total Ankle Replacement
- Anterior Approach (Active Comparator)
  Interventions: Procedure: Total Ankle Replacement

INTERVENTIONS:
Procedure: Total Ankle Replacement — Participants will undergo either lateral approach or anterior approach when having a total ankle replacement

SUMMARY:
A minimum of 50 patients with ankle end-stage arthritis will be randomized in two parallel groups for surgery. One group will receive a total ankle replacement through an anterior approach and the other group a total ankle replacement via a lateral approach. Patients will be evaluated for a mean follow-up of two years in terms of complications, implant survival and functional results. One of the primary objectives of the study is analyzing the safety of the lateral and anterior approaches for total ankle replacement.

DETAILED DESCRIPTION:
A minimum of 50 patients with ankle end-stage arthritis will be randomized in two parallel groups for surgery. One group will receive a total ankle replacement through an anterior approach and the other group a total ankle replacement via a lateral approach. Patients will be evaluated for a mean follow-up of two years in terms of complications, implant survival and functional results. One of the primary objectives of the study is analyzing the safety of the lateral and anterior approaches for total ankle replacement.

The anterior approach uses an interval between the anterior tibial tendon and the extensor digitorum longus tendon to reach the joint. The anterior tibial artery and the deep peroneal nerve must be identified and protected. Once the ankle is reached, the joint is roughly prepared and the cutting guides for the implants are inserted. The position is checked, and the size of the prosthesis is determined. There are several commercial prostheses designed for this approach, although we decided to use the Infinity™ Total Ankle System (Stryker Medical®) to minimize bias. After alignment examination, the implants are inserted, the planes are closed, and the wound is covered. The patient is placed in a cast for three weeks and starts weight-bearing in a boot after this period, using it for three more weeks.

The lateral approach utilizes an incision over the posterior aspect of the fibula. The lateral malleolus is osteotomized 1.5cm proximal to the joint and reflected distally to provide access to the articulation. An external frame is placed around the limb that supplies guidance for the prosthesis cuts. The sizing and position are determined and a Trabecular Metal Total Ankle™ (ZimmerBiomet®) is placed, the only available implant for the lateral approach. The fibula is reduced and fixed using a low profile anatomical lateral plate and screws. Planes are closed, the wound protected, and a cast placed. The post-operative carry is the same as the anterior approach.

Weight bearing CT (WBCT) scans will be used to evaluate outcomes. WBCT is the standard of care for the preoperative and postoperative assessment of patients undergoing total ankle replacement in our institution. Many secondary outcomes will be also evaluated through WBCT since they can better depict alignment, predict failure and diagnose complications (subsidence, cysts). No extra WBCT will be performed other than what we normally do for patients.

Randomization will be performed previously at the beginning of the study and will be performed by an outside researcher. Allocation will happen during surgery scheduling.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must be older than 18 and younger than 90 years of age, both genders.
* Participants must be experiencing symptoms related to their baseline condition for at least six months before the surgery.
* Clinical and radiographical clinical diagnosis of ankle arthritis.
* Surgical planning of total ankle replacement.

Exclusion Criteria:

* Previous surgery for total ankle replacement or ankle arthrodesis.
* History or documented evidence of autoimmune or peripheral vascular diseases.
* History or documented evidence of peripheral neuropathy (nervous compression syndrome, tarsal tunnel syndrome) or systemic inflammatory disease a (rheumatoid arthritis, seronegative, connective, etc.);
* Any condition that represents a contraindication of the proposed therapies.
* Any physical or social limitation that makes the protocol continuation unviable.
* Impossibility or incapacity to sign the informed Consent Form.
* Presence of infectious process (superficial on the skin and cellular tissue, or deep in the bone) in the region to be treated.
* Pregnancy.
* Clinical and imaging diagnosis of untreated osteoporosis.
* Serum vitamin D levels below 20ng/ml.
* Non-palpable anterior or posterior tibial pulse; or abnormal capillary filling.
* Tumor lesions (primary or secondary tumors).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-05 (Estimated); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Complications | 6 months post-surgery
  To compare major and minor complications of patients undergoing TAR through lateral and anterior approaches.
Survival | 6 months post-surgery
  To compare survival rate between the two techniques.

SECONDARY OUTCOMES:
Foot and Ankle Ability Measure | 96 weeks post-surgery
  To compare patient reported outcomes (PROs) between the two groups.
PROMIS Global Health | 96 weeks post-surgery
  To compare patient reported outcomes (PROs) between the two groups.
PROMIS Depression - Short Form | 96 weeks post-surgery
  To compare patient reported outcomes (PROs) between the two groups.
PROMIS Physical Function 8B | 96 weeks post-surgery
  To compare patient reported outcomes (PROs) between the two groups.
PROMIS Pain Interference 8A | 96 weeks post-surgery
  To compare patient reported outcomes (PROs) between the two groups.
Pain VAS Scale | 96 weeks post-surgery
  To compare patient reported outcomes (PROs) between the two groups.
Tampa Scale for Kinesiophobia | 96 weeks post-surgery
  To compare patient reported outcomes (PROs) between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: John Femino, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No